CLINICAL TRIAL: NCT03061669
Title: Respiratory Monitoring During Right Heart Catheterization to Differentiate Between Various Types of Pulmonary Hypertension; The Effects of the Cardiovascular System on the Lung Mechanical Properties
Brief Title: Respiratory Monitoring During Right Heart
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Technion, Israel Institute of Technology (Other)
Responsible Party: Principal Investigator, yair feld MD, Principal investigator, Rambam Health Care Campus
Other Study IDs: 0370-16
Record Dates: First submitted 2017-02-03; First posted 2017-02-23 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Pulmonary Hypertension; Heart Failure
Keywords: heart failure; pulmonary hypertension; right heart catheterization
MeSH Terms: conditions — Hypertension, Pulmonary; Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Respiratory monitoring during right heart catheterization to differentiate between various types of pulmonary hypertension; The effects of the cardiovascular system on the lung mechanical properties.

DETAILED DESCRIPTION:
Differentiation between different kinds of pulmonary hypertension (PHTN) requires right heart catheterization. Monitoring heart failure patients is challenging in many. The study will enroll patients undergoing right heart catheterization (RHC) for the evaluation of heart failure and PHTN, based on the regular clinical practice. The regular indices as the right ventricle pressure (RVP), pulmonary artery pressure (PAP), pulmonary artery wedge pressure (PAWP), and cardiac output will be measured with the Swan Ganz Catheter and recorded.

Noninvasive measurement of the respiratory flow will be acquired by a medical approved flow-meter that is mounted on a simple plastic breathing mask.

Non-invasive system that includes three accelerometers that are attached to the chest and epigastrium of the patient will be used to measure respiratory chest wall dynamics.

Through evaluating the correlation between the invasive and non-invasive measurements the study intends to prove the ability of the non-invasive system to provide the required information.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing right heart catheterization

Exclusion Criteria:

* Inability or unwillingness to follow or to sign the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing right heart catheterization (RHC) for the evaluation of heart failure and pulmonary hypertension, based on the regular clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-02-26 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Pulmonary artery pressure | only during the procedure of right heart catheterization
  In mmHg measured by Swan-Ganz catheter
Respiratory flow | only during the procedure of right heart catheterization
  ml units
Chest wall acceleration | only during the procedure of right heart catheterization
  local tidal displacement

SECONDARY OUTCOMES:
Right ventricle pressure | only during the procedure of right heart catheterization
  In mmHg measured by Swan-Ganz catheter
Pulmonary artery wedge pressure | only during the procedure of right heart catheterization
  In mmHg measured by Swan-Ganz catheter

CONTACTS AND LOCATIONS:
Overall Officials: Yair Feld, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam medical center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No